CLINICAL TRIAL: NCT04617951
Title: Effect of Ishige Okamurae Extract on Musculoskeletal Biomarkers in Adults With Relative Sarcopenia: a Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Effect of Ishige Okamurae Extract on Musculoskeletal Biomarkers in Adults With Relative Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-2020-029
Record Dates: First submitted 2020-10-23; First posted 2020-11-05 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ishige Okamurae extracts group (Experimental): This group takes Ishige Okamurae extracts for 12 weeks.
  Interventions: Dietary Supplement: Ishige Okamurae extracts group
- Placebo group (Placebo Comparator): This group takes placebo for 12 weeks.
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Ishige Okamurae extracts group — Ishige Okamurae extracts 300 mg/day for 12 weeks
  Arms: Ishige Okamurae extracts group
Dietary Supplement: Placebo group — Placebo 300 mg/day for 12 weeks
  Arms: Placebo group

SUMMARY:
The investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of Ishige Okamurae extracts on muscle strength, muscle mass, and muscle function in adults with relative sarcopenia for 12 weeks.

DETAILED DESCRIPTION:
A previous study has indicated that Ishige Okamurae extracts may increase muscle mass and strength. Therefore, the investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of Ishige Okamurae extracts on muscle strength, muscle mass, and muscle function in adults with relative sarcopenia; the safety of the compound are also evaluated. The Investigators examine the peak torque/body weight at 60°/s knee extension, handgrip strength, skeletal muscle mass, physical performance, and metabolic parameters at baseline, as well as after 6 and 12 weeks of intervention. Eighty adults were administered either 300 mg of Ishige Okamurae extracts or a placebo each day for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* <110% of the standard lean body mass as measured using the body composition analyzer
* Body mass index (BMI) ranging from 18.5 to 30.0 kg/m2
* Those who have an average protein intake of 60 g or more/day.

Exclusion Criteria:

* Abnormal liver or renal function (more than twice the normal upper limit of the research institute)
* Uncontrolled diabetes mellitus (>160 mg/dL of fasting blood sugar)
* History of fracture during the previous year
* Uncontrolled hypertension (>160/100 mmHg)
* Uncontrolled thyroid diseases.
* History of serious cerebro-cardiovascular diseases or cancer such as angina or myocardial infarction within 6 months
* History of any central bone fracture within 1 year
* History of medication for psychiatric diseases such as severe depression, schizophrenia, drug intoxication.
* Alcohol abuser
* Allergic reaction to Ishige Okamurae
* Those who participated in other drug clinical trials within 1 month from the screening date.
* Severe gastrointestinal symptoms such as heartburn and indigestion
* Those who are pregnant, lactating, or plan to become pregnant during the clinical trial
* Those who are judged to be unsuitable by the PI for other reasons

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
muscle strength | 12 weeks
  the peak torque at 60°/s knee extension (/kg)

SECONDARY OUTCOMES:
appendicular skeletal mass/(height x height) | 12 weeks
  using dual-energy X-ray absorptiometry measured at baseline and after 12 weeks
appendicular skeletal mass/weight x 100 | 12 weeks
  using dual-energy X-ray absorptiometry measured at baseline and after 12 weeks
skeletal Muscle Mass Index/(height x height) | 12 weeks
  using dual-energy X-ray absorptiometry measured at baseline and after 12 weeks
concentration of creatinine kinase (IU/L) | 12 weeks
  creatinine kinase (IU/L) measured at baseline and after 12 weeks
concentration of lactate (mg/dL) | 12 weeks
  lactate (IU/L) measured at baseline and after 12 weeks
EuroQol five dimensional three levels | 12 weeks
  an index of life quality, minimum, maximum values (-0.171, 1), higher scores mean a better outcome, which will be measured at baseline and after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeungsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SR, Lee YL, Lee SY. Effect of Ishige okamurae extract on musculoskeletal biomarkers in adults with relative sarcopenia: Study protocol for a randomized double-blind placebo-controlled trial. Front Nutr. 2022 Sep 27;9:1015351. doi: 10.3389/fnut.2022.1015351. eCollection 2022. PMID 36238450